CLINICAL TRIAL: NCT02818023
Title: Dose-seeking Study of Pembrolizumab Plus Vemurafenib and Cobimetinib for Therapy of Advanced Melanoma
Brief Title: Dose-seeking Study of Pembrolizumab Plus Vemurafenib and Cobimetinib Advanced Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Accrual to trial stopped due to high toxicity even at lowest dose of combination treatment. Patients on trial tolerating treatment at time of accrual closure still continued to receive treatment.
Sponsor: Yana Najjar (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Yana Najjar, Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-131
Record Dates: First submitted 2016-06-07; First posted 2016-06-29 (Estimated); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab; Vemurafenib; cobimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pembrolizumab plus vemurafenib and Cobimetinib (Experimental): * Pembrolizumab will be given at a dose of 200 mg q3 weeks (this is the standard dosage, ), and vemurafenib/cobimetinib will be given at 480 mg twice daily/20 mg daily, 720 mg twice daily/40 mg daily, or 960 mg twice daily/60 mg daily. Treatment with pembrolizumab and vemurafenib will commence on the same day.
  * One cycle of treatment will be defined as one dose of pembrolizumab and 3 weeks of vemurafenib.
  Interventions: Drug: Pembrolizumab; Drug: Vemurafenib; Drug: Cobimetinib

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab will be given at a dose of 200 mg q3 weeks (this is the standard dosage, ). Treatment with pembrolizumab and vemurafenib will commence on the same day.
  One cycle of treatment will be defined as one dose of pembrolizumab and 3 weeks of vemurafenib.
Drug: Vemurafenib — Vemurafenib will be given at 480 mg twice daily, 720 mg twice daily, or 960 mg twice daily. Treatment with pembrolizumab and vemurafenib will commence on the same day.
  One cycle of treatment will be defined as one dose of pembrolizumab and 3 weeks of vemurafenib.
Drug: Cobimetinib — Cobimetinib will be given at 20 mg once daily, 40 mg once daily, or 60 mg once daily. Treatment with cobimetinib will commence on the same day. Cobimetinib will be given daily for 21 days, then held for 7 days.

SUMMARY:
The study plans to treat patients with pembrolizumab and thus blocking the PD-1/PD-L1 axis would render tumor-infiltrating lymphocytes (TILs) in the tumor parenchyma more functional as a consequence of BRAF inhibition, such that T cell activation by BRAFi would not be dampened by the PD-1/PD-L1 interaction. This combination would reverse dysfunction among T cells in the tumor parenchyma, maximizing T cell mediated immune anti-tumor efficacy. Progression free survival (PFS) with pembrolizumab in KEYNOTE-001 was 57% at 6 months, and 46.4% in the more recently reported phase III trial. PFS with vemurafenib treatment in BRIM-3 was ~50% at 6 months. Combined treatment with pembrolizumab, cobimetinib and vemurafenib for BRAF mutant melanoma is hypothesized to be safe and to improve the PFS compared to these recent historical controls. Because this combination has not yet been tested, and because the primary objective is to assess safety, the investigators are staging accrual in the first phase of the trial. The study aims to accrue up to 30 patients to the mTPI design of this study with the expectation that there will be at least 30 patients treated at RP2D. In case there are less than 30 patients on the RP2D, additional patients will be accrued. Patients will continue to receive treatment with pembrolizumab, vemurafenib and cobimetinib until disease progression or dose limiting toxicity. Patients with treatment response and no dose limiting toxicity may receive treatment with pembrolizumab for up to 24 months.

DETAILED DESCRIPTION:
Pembrolizumab will be given at a dose of 200 mg q3 weeks (this is the standard dosage, ), and vemurafenib/cobimetinib will be given at 480 mg twice daily/20 mg daily, 720 mg twice daily/40 mg daily, or 960 mg twice daily/60 mg daily. Treatment with pembrolizumab, vemurafenib and cobimetinib will commence on the same day.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent obtained prior to the initiation of study procedures.
2. Male and female subjects who are at least 18 years of age.
3. Histologically confirmed unresectable stage III or stage IV melanoma (AJCC 7th edition classification). Cutaneous melanoma and mucosal melanoma will be eligible.
4. Only patients with BRAF V600E or V600K mutated tumors will be enrolled.
5. Baseline skin exam is required for all patients. Note: Cutaneous squamous cell carcinoma (SCC) lesions identified at baseline must be excised.
6. Measurable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST v1.1). Baseline measurements must be obtained within 4 weeks prior to registration.
7. Adequate hematologic, renal, and liver function as evidenced by the following (within 4 weeks prior to starting the study drugs):

   * WBC ≥ 3,000/mm3
   * ANC ≥ 1500
   * Hemoglobin ≥ 9g/dL (women) or ≥ 11g/dL (men) Platelets ≥ 100,000/mm3 Serum Creatinine ≤ 1.5 x upper limit of normal (ULN)
   * Serum Bilirubin ≤ 1.5 x ULN
   * Serum AST and ALT ≤ 2.5 x ULN

   Note: (supportive transfusions will be allowed during screening and during treatment as deemed necessary by the treating physician)
8. EKG documenting QTc interval < 480 msec and no clinically significant arrhythmia
9. Fully recovered from any effects of major surgery, and be free of significant infection.
10. ECOG performance status of 0 or 1.
11. Female patients of child bearing potential must have a negative pregnancy test within 7 days from the time of registration .
12. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
13. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for greater than 1 year.
14. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
15. Patients with brain metastases may be enrolled if brain metastases have been treated by surgery and/or radiation and are stable on 2 week repeat scan.

Exclusion Criteria:

1. Serious clinically significant illnesses, such as: cardiovascular disease (uncontrolled congestive heart failure, uncontrolled hypertension, cardiac ischemia, myocardial infarction, and severe cardiac arrhythmia), bleeding disorders, symptomatic autoimmune diseases (such as inflammatory bowel disease, autoimmune hepatitis, uncontrolled hypo or hyperthyroidism), severe obstructive or restrictive pulmonary diseases, retinopathy, active systemic infections, and inflammatory bowel disorders.
2. Known HIV or AIDS-related illness, or active HBV and HCV.
3. Has a known history of active TB (Bacillus Tuberculosis)
4. History of grade 4 immune-related adverse events requiring treatment with prednisone, or grade 3 immune-related adverse events requiring prednisone >10 mg/kg for >12 weeks, if previously treated with ipilimumab.
5. Prior therapy with anti-PD-1 agent(s) in the metastatic setting. Treatment with anti-PD1 in the adjuvant setting is permitted.
6. Prior therapy with a BRAF and/or MEK and/or ERK inhibitors in the metastatic setting. Treatment with BRAF/MEKi in the adjuvant setting is permitted.
7. Refractory nausea, vomiting, small bowel resection or any other gastrointestinal ailment that would preclude study drug absorption.
8. Cardiac abnormalities

   * Mean QTc interval ≥ 480 msec at screening.
   * ACS/AMI -within 24 weeks prior to screening.
   * PCI/PTCA -within 24 weeks prior to screening.
   * Symptomatic heart failure - NYHA Class ≥ II symptoms.
9. Active infection within one-week prior to study, including unexplained fever
10. Systemic steroid or other immunosuppressive therapy within 4 weeks of starting the study.
11. Lactating females and/or pregnant females.
12. Any significant psychiatric disease, medical or other condition, which in the opinion of the principal investigator could prevent adequate informed consent or compromise participation in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-07-13 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Percentage of participants that experience a dose-limiting toxicity | Up to 2 years
  determine the safety and maximum tolerated dose of vemurafenib and cobimetinib with pembrolizumab

SECONDARY OUTCOMES:
overall response rate (ORR) | Up to 2 years
progression free survival | Up to 2 years
overall survival | up to 2 years

OTHER OUTCOMES:
assessment of tumor microenvironment and immune response via biomarker level measurement | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yana M. Najjar, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Cancer Center Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No